CLINICAL TRIAL: NCT01829594
Title: Case Managers to Frail Older People a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Jimmie Kristensson, PhD, Senior Lecturer, Lund University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 499/2008
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Frail Elderly
Keywords: Case Management; Frail Elderly; Health Services Administration; Delivery of Health Care; Accidental Falls; Health Status; Health Care Economics
MeSH Terms: interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Case Management (Experimental)
  Interventions: Other: Case management

INTERVENTIONS:
Other: Case management — Nurses and a physiotherapist (PT) worked as case managers (CM). The intervention lasted 12 months and comprised 4 dimensions. The first was traditional CM tasks: assessment, planning, monitoring, care coordination and evaluation. Home visits were made at least once a month. The second and third was general and specific information related to the participants' situation. The fourth part included aspects of continuity and safety. The PT also paid home visits and made an assessment regarding physical function and balance. The intervention consisted of multidimensional prevention of falls and/or consequences of falls, and supporting and motivating the participant to increased physical activity. When those in the control group had participated for 12 months they were offered the intervention.

SUMMARY:
The aim of is to test the effects of a model for care (case management) to older people with high healthcare consumption and functional dependency on healthcare consumption, quality of life, functional ability and experiences of care.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 or over
* need help with at least two activities of daily living
* been admitted to hospital on at least two occasions, or
* have had at least four contacts with outpatient or primary care during the previous twelve months,
* be able to communicate verbally
* have no cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 153 (Actual)
Dates: Start 2006-10; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Health care consumption | two years (one year before vs after baseline)
Health care costs | two years (one year before vs after baseline)
Feelings of loneliness | baseline and then after 3,6,9,12,24 months
Depressive symptoms | baseline and then after 3,6,9,12,24 months
Health Related Quality of Life | baseline and then after 3,6,9,12,24 months
Number of falls | baseline and then after 3,6,9,12,24 months

SECONDARY OUTCOMES:
Life Satisfaction | baseline and then after 6,12,24 months
Health complaints | baseline and then after 3,6,9,12,24 months
Knowledge about prescribed drugs | baseline and then after 3,6,9,12,24 months
Attitudes towards prescribed drugs | baseline and then after 3,6,9,12,24 months
Drug use | baseline and then after 3,6,9,12,24 months
Activities and social participation | baseline and then after 3,6,9,12,24 months
Functional capacity | baseline and then after 3,6,9,12,24 months
Balance | baseline and then after 3,6,9,12,24 months
Timed up and go (TUG) | baseline and then after 3,6,9,12,24 months
Risk of falling | baseline and then after 3,6,9,12,24 months
Fear of Falling | baseline and then after 3,6,9,12,24 months

OTHER OUTCOMES:
Experiences of care | approximately one year
  qualitative interviews with participants, next of kins and case managers

CONTACTS AND LOCATIONS:
Overall Officials: Ingalill Rahm Hallberg, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Faculty of Medicine, Department of Health Sciences, Lund, Sweden

REFERENCES:
- [Result] Kristensson J, Ekwall AK, Jakobsson U, Midlov P, Hallberg IR. Case managers for frail older people: a randomised controlled pilot study. Scand J Caring Sci. 2010 Dec;24(4):755-63. doi: 10.1111/j.1471-6712.2010.00773.x. PMID 20409057